CLINICAL TRIAL: NCT05749458
Title: Retrospective Study on Maternal and Neonatal Risk Factors That Contribute to Hypoxic Ischemic Encephalopathy in Neonates
Brief Title: Maternal and Neonatal Risk Factors of HIE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Mamdouh Kemaly, Resident, Assiut University
Other Study IDs: Risk factors in HIE neonates
Record Dates: First submitted 2023-01-31; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Hypoxic Ischemic Encephalopathy of Newborn

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The current work aims to:

The primary aim in this study was to identify the contribution of maternal, pregnancy, birth and neonatal factors to encephalopathic features in new born infants.

The secondary aim of this study is to reduce the burden on the country by decreasing the rate of neonatal encephalopathy, decreasing the different grades of neurodevelopmental impairment and improvement the quality of life.

DETAILED DESCRIPTION:
Brain injury in the full-term and near-term gestation neonate is a significant contributor to mortality and long-term morbidity, secondary to the vulnerability of the developing brain to injury. Causes of early brain injury include stroke, birth trauma, metabolic or genetic disorders, neonatal-onset epilepsies, and a variety of perinatal events that lead to decreased blood flow or oxygen delivery to the brain. This last cause is the most common cause of perinatal brain injury. It usually presents with neonatal encephalopathy, or an abnormal neurological examination and is estimated to occur in 3 to 5 in 1000 live births.

The Sarnat and Sarnat classification is still the universally accepted scoring system to provide information about the prognosis for the asphyxiated neonate. This staging is based on the infant's clinical presentation, examination findings and the presence of seizures, with emphasis on the duration of symptoms.

Martinez-Biarge et al. reported some intrapartum factors associated with the development of HIE- Intrapartum maternal fever, prolonged rupture of membranes, Placental abruption, Ruptured uterus, thick meconium, and gestational age ≥ 41 weeks. In their case-control study of infants born beyond 36 weeks gestation, Hayes et al. identified several risk factors for the development of HIE including thick meconium, fetal growth restriction, large head circumference, oligohydramnios, male fetal sex, fetal bradycardia, maternal pyrexia, and increased uterine contractility. Previously identified antenatal risk factors for HIE include nulliparity, gestation > 41 weeks, intrauterine growth restriction, maternal age > 35 years, and urinary tract infection during pregnancy. Previously identified intrapartum risk factors for HIE include sentinel events, emergency cesarean delivery, prolonged rupture of membranes, presence of meconium, shoulder dystocia, maternal fever, and clinical chorioamnionitis.

Also, associated factors of HIE include maternal factors such as maternal age (years), parity (primigravida- multigravida), maternal hypertension, pre-eclampsia, gestational DM, Previous fetal death/stillbirth and prior cesarean section. maternal pre-eclampsia with HELLP syndrome and umbilical cord prolapse have been shown to be a risk for asphyxia (14). Route of delivery (Vaginal - Cesarean section) and neonatal factors as gestational age (weeks), gender, Birth weight (grams) and Apgar score if available. An Apgar scores at 5 min provides useful prognostic data before other evaluations are available. Low Apgar scores at 1, 5 and 10 min have been found to be markers with possible increased risk of death or chronic motor disability.

ELIGIBILITY:
Inclusion Criteria:

* all neonates less than 28 days old newborns, who were admitted to the Neonatal intensive care Unit Assiut University Children's Hospital, from January 2019 till the end of December 2023.

Exclusion Criteria:

* Those newborn infants with stillbirth, congenital anomaly, and chromosomal abnormalities or infants with microbiological evidence of early neonatal infection were excluded from the study.

Ages: 1 Day to 28 Days | Sex: All
Age Groups: Child
Study Population: the study population: all neonates less than 28 days old newborns, who were admitted to the Neonatal intensive care Unit Assiut University Children's Hospital, from January 2019 till the end of December 2023.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Identify the contribution of maternal, pregnancy, birth and neonatal factors to increase incidence of encephalopathic features in new born infants. | Baseline
  retrospective study of newborns, who were admitted to the Neonatal intensive care Unit Assiut University Children's Hospital, from January 2019 till the end of December 2023.All outcome measures were summarized using frequencies and percentages or means ± standard deviations, stratified by group (HIE group vs. Non-HIE group).
  The categorical data were analyzed for statistical significance (p < 0.05) by Chi-square test or Fisher exact test, or Student t-test. The odds ratio and 95% CI were calculated for those with statistical significance. Stepwise multiple logistic regression analysis used to determine the independent factors that may predispose an infant to HIE.

CONTACTS AND LOCATIONS:
Overall Officials: Abdellatif M. Abd-Elmoaz, Professor, Study Director — Assiut University; Mohamed G. Abo-Elela, Professor, Study Director — Assiut University

REFERENCES:
- [Background] Martinez-Biarge M, Diez-Sebastian J, Wusthoff CJ, Mercuri E, Cowan FM. Antepartum and intrapartum factors preceding neonatal hypoxic-ischemic encephalopathy. Pediatrics. 2013 Oct;132(4):e952-9. doi: 10.1542/peds.2013-0511. Epub 2013 Sep 9. PMID 24019409
- [Background] Peebles PJ, Duello TM, Eickhoff JC, McAdams RM. Antenatal and intrapartum risk factors for neonatal hypoxic ischemic encephalopathy. J Perinatol. 2020 Jan;40(1):63-69. doi: 10.1038/s41372-019-0531-6. Epub 2019 Oct 14. PMID 31611618
- [Background] Parker SJ, Kuzniewicz M, Niki H, Wu YW. Antenatal and Intrapartum Risk Factors for Hypoxic-Ischemic Encephalopathy in a US Birth Cohort. J Pediatr. 2018 Dec;203:163-169. doi: 10.1016/j.jpeds.2018.08.028. Epub 2018 Sep 27. PMID 30270166
- [Background] Torbenson VE, Tolcher MC, Nesbitt KM, Colby CE, El-Nashar SA, Gostout BS, Weaver AL, Mc Gree ME, Famuyide AO. Intrapartum factors associated with neonatal hypoxic ischemic encephalopathy: a case-controlled study. BMC Pregnancy Childbirth. 2017 Dec 11;17(1):415. doi: 10.1186/s12884-017-1610-3. PMID 29228911